CLINICAL TRIAL: NCT07373964
Title: A Prospective, Single-Arm, Single-Center Phase II Study Evaluating the Efficacy and Safety of Chidamide Tablets Combined With PD-L1 Inhibitor, Carboplatin, and Etoposide as First-Line Treatment in Patients With Extensive-Stage Small-Cell Lung Cancer (ES-SCLC)
Brief Title: A Prospective, Single-Arm, Single-Center Phase II Study Evaluating the Efficacy and Safety of Chidamide Combined With PD-L1 Inhibitor, Carboplatin, and Etoposide as First-Line Treatment in Patients With Extensive-Stage Small-Cell Lung Cancer (ES-SCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q115
Record Dates: First submitted 2026-01-21; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: Chidamide Tablets； PD-L1 Inhibitor (as per chosen drug's prescribing information)；Carboplatin； Etoposide

INTERVENTIONS:
Drug: Chidamide Tablets； PD-L1 Inhibitor (as per chosen drug's prescribing information)；Carboplatin； Etoposide — Induction Phase: Chidamide 15 mg orally on days 1, 4, 8, 11, 15, and 18 of each 21-day cycle for 4 cycles.PD-L1 inhibitor, carboplatin, and etoposide are administered per their respective prescribing information.
  Maintenance Phase: Chidamide 20 mg orally twice weekly (at least 3 days apart) until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.PD-L1 inhibitor is administered per their respective prescribing information.

SUMMARY:
This is a Phase II, single-arm, single-center study evaluating Chidamide combined with a PD-L1 inhibitor, carboplatin, and etoposide as first-line therapy in extensive-stage small-cell lung cancer (ES-SCLC) patients. The primary objective is to assess Progression-Free Survival (PFS) per RECIST v1.1. Secondary objectives include Objective Response Rate (ORR), Disease Control Rate (DCR), Duration of Response (DOR), Overall Survival (OS), and safety. Approximately 36 participants will receive induction therapy (Chidamide + chemotherapy + PD-L1 inhibitor) for 4 cycles, followed by Chidamide maintenance until progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years.
* Histologically confirmed ES-SCLC, unsuitable for local radical therapy.
* No prior systemic therapy for ES-SCLC.
* ECOG performance status 0-1.
* At least one measurable lesion per RECIST v1.1.
* Expected survival ≥3 months.
* Adequate organ function (hematological, hepatic, renal, cardiac).
* Effective contraception from consent until 180 days after last dose.
* For active HBV infection: HBV DNA <2000 IU/mL within 28 days before treatment and on stable antiviral therapy.
* Recovery from prior therapy toxicities to ≤ Grade 1 (except alopecia).
* Signed informed consent.

Exclusion Criteria:

* Factors significantly affecting oral drug absorption.
* Prior HDAC inhibitor or immune checkpoint inhibitor therapy.
* Known allergy to any study drug component.
* Other malignancy within past 5 years (except certain cured cancers).
* Participation in another clinical trial within 4 weeks.
* Immunodeficiency, HIV positivity, or organ transplant history.
* Uncontrolled cardiovascular disease or QTc >450 ms.
* Pregnancy, lactation, or unwillingness to use effective contraception.
* Other severe comorbid conditions deemed unsafe by investigator.
* History of neurological or psychiatric disorders.
* Any condition making the patient unsuitable per investigator judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2027-10-14 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) per RECIST v1.1 as assessed by the investigator. | baseline up to approximately 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST v1.1. | baseline up to approximately 24 months
Disease Control Rate (DCR) per RECIST v1.1. | baseline up to approximately 24 months
Duration of Response (DOR) per RECIST v1.1 | baseline up to approximately 24 months
Overall Survival (OS) | baseline up to approximately 24 months
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | baseline up to approximately 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China